CLINICAL TRIAL: NCT06768593
Title: Evaluation of the Effectiveness of Ultrasound-Guided Recto-Intercostal Fascial Plane (RIFP) Block in Postoperative Analgesia Management in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Recto-Intercostal Fascial Plane (RIFP) Block in Laparoscopic Cholecystectomy Patients
Acronym: RIFPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assist Prof, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 4
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Cholecystectomy; Pain Management; Plane Block; Acute Pain
Keywords: pain management; Recto-Intercostal Fascial Plane (RIFP) Block; laparoscopic cholecystectomy
MeSH Terms: conditions — Agnosia; Acute Pain; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification II-III, scheduled for laparoscopic cholecystectomy operation will be included in the study. Patients will be randomly divided into two groups (Group R=RIFP block group, Group K = control group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcomes assessor and participants will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R = RIFP Block group (Experimental): RIFP block will be performed and standard postoperative pain management protocols will be applied.
  Interventions: Procedure: RIFP Block; Other: Postoperative pain management
- Group K = Control group (Active Comparator): Standard postoperative pain management protocols will be applied. No plane block will be applied.
  Interventions: Other: Postoperative pain management

INTERVENTIONS:
Procedure: RIFP Block — After aseptic conditions are ensured, with high-frequency linear US probe (11-12 MHz, Vivid Q) and a 22-G 80-mm needle (Pajunk Sonoplex Nanoline Stim Cannula, Germany) bilateral block will be applied to Group R. As the patient is in supine position, the USG probe is placed in transverse plane on the sternum and will be directed downwards and laterally and rotated to determine the xiphoid and just below the rectus abdominis muscles. Costal cartilage and rectus abdominis muscle sonographically will be shown. This region corresponds to the 3-4 cm lateral and 3-4 cm caudal region of the xiphoid. Using the in-plane technique, the block needle will be advanced in the caudal-cephalic direction, and 5 ml saline will be injected into the area between the rectus muscle and costal cartilage to verify the block location. 30 ml of 0.25% bupivacaine (Buvacaine, Polifarma ®) will be injected to each side, which corresponds to 60 ml total local anesthetic-saline mixture in Group R.
  Arms: Group R = RIFP Block group
Other: Postoperative pain management — Ibuprofen 400 mg (Ibuprofen, Polifarma ®) and tramadol 100 mg (Contramal, Abdi İbrahim ®) IV single bolus dose will be given 20 minutes before the end of the surgical procedure for postoperative analgesia.
  NRS scores at rest and while moving will be evaluated and recorded and if the NRS score is ≥ 4, meperidine 0,5 mg/kg (Aldolan®) IV will be administered as a rescue analgesic.

SUMMARY:
Ultrasound-guided Recto-Intercostal Fascial Plane (RIFP) Block is performed by injecting local anesthetic deep between the 7th rib and the costochondral aspect of the rectus muscle. It provides blockage of both the anterior and lateral cutaneous branches of T6-T10/11 and analgesia of the sternum, epigastrium, and upper abdomen (1).

Studies show that RIFP block is effective for postoperative analgesia, sternum revision, and cardiac surgery. However, its effect on patients undergoing laparoscopic cholecystectomies has not been studied yet. The investigators hypothesize that RIFP block performed in laparoscopic cholecystectomies would reduce postoperative rescue analgesic use and postoperative opioid consumption in the first 24 hours after surgery.

DETAILED DESCRIPTION:
Cholecystectomy is the most common abdominal surgical procedure performed in developed countries and is usually performed laparoscopically. Many factors play a role in the pain that develops after laparoscopic cholecystectomy and it has both somatic and visceral components. Phrenic nerve irritation as a result of CO₂ insufflation into the peritoneal cavity, abdominal distension, tissue trauma, trauma due to gallbladder removal, sociocultural differences, and individual factors are the factors that play a role in the emergence of this pain. Postoperative pain is an acute pain that is accompanied by an inflammatory process that occurs due to surgical trauma and gradually decreases with tissue healing. Pain in the postoperative period in patients undergoing laparoscopic cholecystectomy is a serious problem that reduces patient comfort and delays the patient's return to normal life after surgery. Effective postoperative pain management prevents many effects such as shallow breathing and delayed mobilization.

RIFPB performed with ultrasound (US) guidance is a new abdominal plane block. The rectus muscle attaches to the cartilage of the 7th rib in the epigastrium on the cranial side. Injecting local anesthetic between the 7th rib and the rectus muscle provides effective analgesia in the sternal, epigastric, and upper abdominal areas. It can be used as a complementary block for thorax, and a stand-alone technique for the abdomen. RIFPB provides analgesia at T6-T10/11 dermatome levels for lateral and medial cutaneous branches. Visualizing son anatomy with US is easy and the spread of local anesthetic can be easily detected. According to the literature, there are case series reporting RIFPB to be effective in cardiac surgery, and sternum revision surgery, both for postoperative analgesia management and as a sole anesthetic method alone. The investigators hypothesize that this block can provide effective postoperative analgesia in laparoscopic cholecystectomy operations due to its mechanism of action. This study aims to evaluate the effectiveness of USG-guided RIFB block for primary postoperative analgesia management after laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II patients
* Laparoscopic cholecystectomy operation under general anesthesia

Exclusion Criteria: patients with

* with a history of bleeding diathesis
* v receiving anticoagulant treatment,
* with allergies or sensitivity to drugs used,
* with an infection on the puncture site
* with a history of alcohol or drug addiction,
* with congestive heart failure
* with liver or kidney disease
* who do not accept the procedure or participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Rescue analgesic use | Need for rescue analgesics at 1, 3, 6, 12,18, and 24 hours postoperatively.
  The primary aim is to investigate postoperative rescue analgesic use and postoperative opioid consumption.

SECONDARY OUTCOMES:
Compare postoperative pain scores (Numeric Rating Scale - NRS scores) | NRS scores at rest and while moving will be evaluated and recorded at 1, 3, 6, 12,18, and 24 hours postoperatively.
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginabl. Higher pain scores mean worse outcome.
  NRS scores at rest and while moving will be evaluated and recorded.
Side effects and complications | Side effects and complications will be evaluated and recorded at 1, 3, 6, 12,18, and 24 hours postoperatively
  Side effects such as nausea, vomiting, sedations, and complications (hematoma, pneumothorax, etc.) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Mega Hospital Complex, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data (IPD).

REFERENCES:
- [Result] Dost B, Turunc E, Ozdemir E. Subxiphoid Pericardial Window Using a Combination of Rectointercostal Fascial Plane Block and Superficial Parasternal Intercostal Plane Block. J Cardiothorac Vasc Anesth. 2024 May;38(5):1282-1283. doi: 10.1053/j.jvca.2024.02.002. Epub 2024 Feb 4. No abstract available. PMID 38453556
- [Result] Ciftci B, Omur B, Alver S, Akin AN, Yildiz Y, Tulgar S. The Medipol Combination: Novel Rectointercostal Fascial Plane Block and Pectointercostal Fascial Plane Block for Postoperative Analgesia Management After Cardiac Surgery: A Report of 15 Cases. A A Pract. 2024 Jun 5;18(6):e01794. doi: 10.1213/XAA.0000000000001794. eCollection 2024 Jun 1. PMID 38836555
- [Result] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Alver S, Sakul BU, Ansen G, Pence KB, Alici HA. Recto-intercostal fascial plane block: Another novel fascial plane block. J Clin Anesth. 2023 Oct;89:111163. doi: 10.1016/j.jclinane.2023.111163. Epub 2023 Jun 7. No abstract available. PMID 37295124